CLINICAL TRIAL: NCT01327924
Title: Ease of Use and Tolerability of Norditropin NordiFlex® in Growth Hormone naïve Children: Impact on Daily Life
Brief Title: Usability and Tolerability of the Norditropin NordiFlex® Injection Device in Children Never Previously Treated With Growth Hormone
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: GH-3870; U1111-1119-8619 (Other: WHO)
Record Dates: First submitted 2011-03-31; First posted 2011-04-04 (Estimated); Last update posted 2014-06-24 (Estimated); Status verified 2014-06

CONDITIONS: Growth Hormone Disorder; Growth Hormone Deficiency in Children; Genetic Disorder; Turner Syndrome; Foetal Growth Problem; Small for Gestational Age; Chronic Kidney Disease; Chronic Renal Insufficiency; Delivery Systems
MeSH Terms: conditions — Genetic Diseases, Inborn; Turner Syndrome; Renal Insufficiency, Chronic | interventions — Growth Hormone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Norditropin NordiFlex® users
  Interventions: Drug: Norditropin NordiFlex®

INTERVENTIONS:
Drug: Norditropin NordiFlex® — Daily administration by subcutaneous injection (under the skin). Starting dose and frequency will be determined by the physician as part of normal clinical practice.

SUMMARY:
This study is conducted in Europe. The purpose of this study is to assess the impact on daily life for children new to using a growth hormone injection device.

ELIGIBILITY:
Inclusion Criteria:

* Growth hormone (GH) treatment naïve subjects for whom it has been decided to initiate GH treatment prior to enrollment into the study
* Subjects who receive Norditropin NordiFlex® according to the SPC

Exclusion Criteria:

* Known or suspected allergy to study product(s) or related products
* Child and/or parent unable to give consent or fill out the questionnaires
* The receipt of any investigational medicinal product within 3 months prior to this study
* Suffer from a life-threatening disease

Max Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Growth hormone treatment naïve children for whom a prescription of Norditropin NordiFlex® is initiated according to the SPC (Summary of Product Characteristics)
Sampling Method: Non-Probability Sample
Enrollment: 77 (Actual)
Dates: Start 2011-04; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Usability of growth hormone injection device assessed by a quantitative scale | after 3 months of growth hormone treatment

SECONDARY OUTCOMES:
Number of adverse events | from 0 - 3 months of growth hormone treatment
Number of technical complaints | from 0 to 3 months of growth hormone treatment

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Paris La Défense Cedex, France

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com